CLINICAL TRIAL: NCT05694780
Title: Sleep Health Care in Pregnancy: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202209036RINC
Record Dates: First submitted 2023-01-05; First posted 2023-01-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Women in the intervention group will receive standard obstetric care plus the STEP intervention which is a 8-week program based on sleep hygiene education and cognitive-behavioral training.
  Interventions: Behavioral: Sleep intervention
- Control (No Intervention): Women in the control group will receive standard obstetric care.

INTERVENTIONS:
Behavioral: Sleep intervention — Standard obstetric care plus the sleep intervention which is a 8-week program based on sleep hygiene education and cognitive-behavioral training.
  Arms: Experimental

SUMMARY:
Sleep disturbances are one of the most frequent complaints brought to the healthcare professionals during routine prenatal care visits.The purpose of this study is to develop and evaluate a Sleep Training and Education Program (STEP) for improving sleep and health in women during pregnancy.

DETAILED DESCRIPTION:
Women in the intervention group will receive standard obstetric care plus the STEP intervention which is a 8-week program based on sleep hygiene education and cognitive-behavioral training.

ELIGIBILITY:
Inclusion Criteria:

* During the first trimester of pregnancy
* Singleton pregnancies

Exclusion Criteria:

* Women have pregnancy-related complications
* Women have diagnosed a psychiatric or sleep disorder

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep by actigraphy | Through study completion, an average of 16 weeks
  Actigraphy is an objective sleep measurement method that assesses physical motion through a small device worn on the non-dominant wrist

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Tsai, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No